CLINICAL TRIAL: NCT00992602
Title: Phase II Study of the Combination of High-Dose Methotrexate and Intrathecal Liposomal Cytarabine in Patients With Leptomeningeal Metastases With or Without Parenchymal Brain Involvement
Brief Title: Liposomal Cytarabine and High-Dose Methotrexate in Treating Patients With Central Nervous System Metastases From Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maciej Mrugala, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6954; NCI-2009-01309 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6954 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Central Nervous System Metastases; Leptomeningeal Metastases; Recurrent Breast Cancer; Stage IV Breast Cancer; Tumors Metastatic to Brain
MeSH Terms: conditions — Meningeal Carcinomatosis; Breast Neoplasms; Brain Neoplasms | interventions — Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (liposomal cytarabine, high-dose methotrexate) (Experimental): See Detailed Description
  Interventions: Drug: methotrexate; Drug: liposomal cytarabine; Other: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: liposomal cytarabine — Given IT or via LP
  Other Names: cytarabine liposome; DepoCyt; DepoCyte; DepoFoam-encapsulated cytarabine; DTC 101
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving liposomal cytarabine and high-dose methotrexate works in treating patients with breast cancer that has spread to the central nervous system. Drugs used in chemotherapy, such as liposomal cytarabine and methotrexate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving liposomal cytarabine with high-dose methotrexate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To show that treatment with high-dose methotrexate (HD-MTX) in combination with intrathecal (IT) sustained-release cytarabine (liposomal cytarabine) will result in median progression-free survival (PFS) greater than 7 weeks for patients with breast cancer and leptomeningeal metastases with or without parenchymal brain involvement.

SECONDARY OBJECTIVES:

I. To describe the overall survival of patients with central nervous system (CNS) metastatic breast cancer treated with the combination of intravenous (IV) HD-MTX and IT Depocyt (liposomal cytarabine).

II. To describe the safety of the combination therapy, in terms of toxicity, adverse events, and the need for dose reductions or schedule modification.

III. To estimate the best overall response rate achieved during treatment with IV HD-MTX and IT Depocyt. Radiographic response will be measured by the Macdonald Criteria using imaging (magnetic resonance imaging [MRI]), and cytologic response will be measured by cerebrospinal fluid (CSF) cytology.

IV. To determine the number of treatment cycles needed to achieve radiographic and cytologic response.

V. To describe response duration in patients who achieve at least partial radiographic response and cytologic clearance.

VI. To define time to clinical progression as measured by Karnofsky performance status (KPS) and neurological exam.

VII. To describe functional status and quality of life of patients, through clinical evaluations of neurological status and patient-reported quality of life (QOL) measured by the Functional Assessment of Chronic Illness Therapy (FACIT) brain and/or CNS questionnaires.

VIII. To correlate response rates with the extent of patient's systemic disease and tumor receptor status (estrogen receptor [ER], progesterone receptor [PR], human epidermal growth factor receptor 2 [Her2]/neu and/or breast cancer, early onset [BRCA] if applicable).

OUTLINE:

INDUCTION THERAPY (WEEKS 1-6): Patients liposomal cytarabine IT or via lumbar puncture (LP) every 14 days beginning in week 1. Patients also receive high-dose methotrexate IV every 14 days beginning in week 2. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY (WEEKS 7-11): Patients achieving complete response (CR), partial response (PR), or stable disease (SD) and CSF negative for malignant cells receive liposomal cytarabine IT or via LP beginning in week 7 and high-dose methotrexate IV beginning in week 8. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY (WEEKS 13-37): Patients achieving CR, PR, or SD and CSF negative for malignant cells receive liposomal cytarabine IT or via LP every 4 weeks beginning in week 13 and high-dose methotrexate IV monthly beginning in week 15. Treatment with liposomal cytarabine repeats every 4 weeks for up to 5 courses and treatment with high-dose methotrexate repeats monthly for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women who are not pregnant (contraception must be used throughout the study)
* Diagnosis of breast cancer with metastases to CNS (regardless of receptor status); leptomeningeal disease must be present with/without parenchymal brain involvement
* Able to provide informed consent
* No prior treatment with whole brain radiotherapy (WBRT); if patient received stereotactic radiosurgery (SRS) prior to enrollment it must be well documented which lesions were treated and untreated index lesions for follow up must be identified; no treatment with SRS will be permitted while on the study; CNS disease must be documented by MRI and CSF cytology
* Karnofsky Performance Status > 60
* White blood cells (WBC) >= 3.0 K
* Absolute neutrophil count (ANC) >= 1.5 K
* Platelets (PLT) >= 100 K
* Hematocrit (HCT) >= 30%
* Glomerular filtration rate (GFR) >= 60 mL/min
* Acceptable liver function (see exclusion criteria)
* Any ongoing therapy for systemic disease allows for the addition of systemic HD-MTX and IT Depocyt; in general patients receiving trastuzumab or lapatinib at the time of enrollment will be allowed to continue; bisphosphonates (i.e., zoledronic acid) and denosumab will be allowed; other non-CNS active chemotherapies might be allowed if no known interactions with study drugs are present; this must be reviewed and approved by the primary investigator on a case-by-case basis
* Mini-mental state examination score of 24 or above

Exclusion Criteria:

* Serum bilirubin > 1.5 x the upper limit of reference range (ULRR)
* Serum creatinine > 1.5 x ULRR or creatinine clearance =< 60 mL/minute (calculated by Cockcroft-Gault formula)
* Potassium, < 3.7 mmol/L despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium out of normal range despite supplementation
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x ULRR
* Alkaline phosphatase (ALP) > 2.5 x ULRR or > 5 x ULRR if judged by the investigator to be related to liver metastases
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Patients with known pleural effusion or ascites
* Prior treatment with whole brain radiotherapy (prior treatment with SRS is allowed under conditions provided in the inclusion criteria)
* Previous allergic or adverse reaction to methotrexate or cytarabine
* Prior treatment with systemic HD-MTX, IT liposomal cytarabine, or IT therapy of any kind
* Prior IT therapy of any kind
* Women who are currently pregnant or breast feeding
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Last dose of prior chemotherapy was less than 4 weeks before the start of study therapy; patients who had no toxicities with prior chemotherapy can start study treatment earlier than 4 weeks
* Stereotactic radiosurgery (SRS) less than 2 weeks before the start of study therapy
* Any unresolved toxicity greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 from previous anti-cancer therapy
* Previous enrollment in the present study
* Major surgery within 4 weeks prior to starting therapy, with the exception of the Ommaya reservoir which can be used for introduction of chemotherapy within 48-72 hours after placement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Mrugala, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Liposomal Cytarabine, High-dose Methotrexate): Induction phase: All patients receive 3 doses of High-Dose Methotrexate (HD-MTX) every 2 weeks given intravenously and 3 doses of Intrathecal (IT) Liposomal Cytarabine (Depocyt) every 2 weeks over 6 weeks.
  Consolidation phase:
  2 additional doses of HD-MTX every 2 weeks and IT-Depocyt every 2 weeks for 4 more weeks.
  Maintenance phase:
  Monthly doses of HD-MTX (up to 6 doses) and IT-Depocyt (up to 5 doses)
  Patients must stop participation anytime MRI shows progressive disease or positive CSF cytology.
Period: Overall Study
Arm/Group | Treatment (Liposomal Cytarabine, High-dose Methotrexate)
Started | 3
Completed | 0
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Liposomal Cytarabine, High-dose Methotrexate)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Survival Free of Neurological Progression, Measured in Weeks
Description: Neurological progression defined by either clinical impression (measured by Karnofsky Performance Status), radiographical response (using Macdonald criteria), or cytologic response (measured by CSF cytology).
Time Frame: Time from start of therapy, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Liposomal Cytarabine, High-dose Methotrexate)
Number analyzed (Participants) | 3
weeks | 6 [-10.7 to 22.7]

2. Secondary Outcome: Overall Survival
Time Frame: Time from start of therapy until death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Liposomal Cytarabine, High-dose Methotrexate)
Number analyzed (Participants) | 3
months | 8.2 [5.5 to 10.9]

ADVERSE EVENTS:
Arm/Group | Treatment (Liposomal Cytarabine, High-dose Methotrexate)
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Liposomal Cytarabine, High-dose Methotrexate) (N=3)
Transaminitis (Hepatobiliary disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Our accrual limitations highlight the challenges of conducting studies in "orphan diseases" such as LC and underscore the importance of multi-center collaboration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No